CLINICAL TRIAL: NCT05336448
Title: POCUS Artificial Intelligence With Portable and Ultraportable Ultrasound Devices in Critically Ill Patients
Brief Title: POCUS AI in Critically Ill Patients
Acronym: PocusAI-Crit
Status: Completed | Type: Observational
Sponsor: Hospital Garcia de Orta (Other)
Responsible Party: Principal Investigator, Filipe André Gonzalez, Senior consultant of Internal Medicine and Intensive Medicine, PhD student, Hospital Garcia de Orta
Other Study IDs: TI 71/2021
Record Dates: First submitted 2022-03-26; First posted 2022-04-20 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective study that aims to assess the differences in point-of-care ultrasound assessment (POCUS) with portable and ultra-portable devices, using conventional vs artificial intelligence (AI) methodologies, performed by experienced vs inexperienced physicians, in critically ill patients.

DETAILED DESCRIPTION:
1. Type of Study Prospective study.
2. Sample Individuals, aged 18 years or over, admitted to the intensive care department, according to the clinical assessment of the medical team, benefit from an ultrasound assessment.

Convenient sample size up to 100 patients

Exclusion criteria:

Patients with atrial fibrillation or other dysrhythmias; Inappropriate acoustic window for ultrasound assessment

c. Devices used The study in question aims to perform an ultrasound using two ultrasound scanners belonging to the Intensive Care Department:

* VenueTM The VenueTM is a portable ultrasound device from GE Healthcare, with touch screen technology, which allows the performance of transthoracic echocardiography and chest ultrasound with M-mode, two-dimensional (2D) and Doppler (color, pulsed, continuous and tissue). Additionally, it uses methodologies that allow the automatic measurement of parameters such as left ventricular ejection fraction, inferior vena cava diameter and its variability, integral time-velocity of flow in the left ventricular outflow tract.
* Butterfly iQ+ The Butterly iQ+ is an ultra-portable ultrasound device, belonging to devices commonly called pocket devices, measuring 163 x 56 x 35 mm. It has a rechargeable battery that allows an autonomy of 2 hours of continuous use. By connecting to a smartphone and after installing the brand application, it allows the performance of transthoracic and pulmonary echocardiography with M-mode, two-dimensional (2D) and color Doppler. It also allows automatic determination of left ventricular ejection fraction. Acquiring images for later review is also possible with this device. d. Variables Demographic, clinical, hemodynamic and respiratory monitoring, laboratory variables - including troponin T, NT-proBNP, creatinine, urea, sodium, potassium, lactate, when available -, severity and mortality scores (SOFA, SAPS- II, APACHE-II) and ultrasound variables. - Echographic variables - transthoracic echocardiography: Acoustic window: nominal qualitative variable, expressed as "good", "reasonable" or "technically difficult". Patient positioning: nominal qualitative variable, expressed in "left lateral decubitus", "right lateral decubitus" or "supine position".

In the 4-chamber apical window (A4C), the following variables should be evaluated (by a physician experienced in echocardiography), with the

Butterfly iQ+ device and then with the VenueTM:

* Left Ventricular Ejection Fraction (LVEF) manual: discrete quantitative variable, expressed in %; refers to the manual measurement of LVEF, obtained through the LV volumes in end-diastole and in end-systole. In the A4C window, the following variables should be evaluated (by a physician experienced in echocardiography and an inexperienced physician), with the Butterfly iQ+ device and then with the VenueTM:
* LVEF auto: discrete quantitative variable, expressed in %; refers to the determination of LVEF through automatic methodology. In the 5-chamber apical window (A5C), the following variables should be evaluated (with the VenueTM device and by a physician experienced in echocardiography):
* Left ventricular outflow tract velocity time integral (LVOT VTI) manual:

discrete quantitative variable, expressed in cm; refers to manual measurement of the LVOT VTI. In the A5C window, the following variables should be evaluated (by a physician experienced in echocardiography and an inexperienced physician), with the VenueTM device:

* LVOT VTI auto: discrete quantitative variable, expressed in cm; refers to the determination of the LVOT VTI through automatic methodology, whose calculation will result from the average of 3 consecutive cycles. In the subcostal window, the following variables should be evaluated (by a physician experienced in echocardiography), with the Butterfly iQ+ device and then with the VenueTM: • Maximum diameter of the manual inferior vena cava (IVC): continuous quantitative variable, expressed in mm, to one decimal place; refers to manual measurement of VCI. • Minimum diameter of manual IVC: continuous quantitative variable, expressed in mm, to one decimal place; refers to manual measurement of VCI. Manual IVC diameter variation: discrete quantitative variable, expressed in %. In the subcostal window, they must be evaluated (by a physician experienced in echocardiography and inexperienced physician), with the

VenueTM device, the following variables:

* Maximum diameter of the inferior vena cava (IVC) auto: continuous quantitative variable, expressed in mm, to one decimal place; refers to the determination of the diameter of the VCI through automatic methodology.
* Minimum diameter of auto VCI: continuous quantitative variable, expressed in mm, to one decimal place; refers to the determination of the diameter of the VCI through automatic methodology.
* Auto IVC diameter variation: discrete quantitative variable, expressed in %. e. Methodology - study stages The ultrasound evaluation of each patient included in the study will be performed by two different doctors. It is intended to evaluate the variables previously discriminated by an experienced doctor in ultrasound and by a non-experienced doctor. Each parameter must be checked in triplicate and registered.

Regarding the echocardiographic assessment, experienced physicians should determine the echographic variables in a conventional way (manual) and also through an automatic methodology, first using the Butterfly iQ+ device and later the VenueTM device. Non-experienced physicians will only perform the determination of variables using the automatic methodology (therefore only the variables for which this option is available). The collection of parameters related to the echocardiographic evaluation will be performed in a previously established order in order to avoid bias in subsequent comparisons. Blood pressure, heart rate, respiratory rate and peripheral oxygen saturation should be recorded during the ultrasound assessment. Regarding laboratory variables, the results available in the analysis of the patient on the day of the ultrasound evaluation will be considered (an additional study will not be requested if any of the measurements has not been previously requested by the attending physician). Any need for vasopressor, inotropic or invasive mechanical ventilation should also be recorded. e) Collection and recording of data Demographic and clinical variables will be collected using the patients' clinical records. The variables referring to the ultrasound assessment will be recorded at the time of their acquisition in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over, admitted to the intensive care department which, according to the clinical assessment of the medical team, would benefit from an ultrasound assessment.

Exclusion Criteria:

* Patients with atrial fibrillation or other dysrhythmias;
* Inappropriate acoustic window for ultrasound assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care department which, according to the clinical assessment of the medical team, would benefit from an ultrasound assessment.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Assess artificial intelligence ultrasound software to assess various echocardiographic variables useful for the management of critically ill patients | up to 48 weeks
  Assess the accuracy of automatic measurements to determine ultrasound parameters using portable versus ultra-portable ultrasound scanners.
  - Assess the accuracy of POCUS performed by inexperienced professionals using portable versus ultraportable ultrasounds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Garcia de Orta, Lisbon, Almada, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varudo R, Gonzalez FA, Leote J, Martins C, Bacariza J, Fernandes A, Michard F. Machine learning for the real-time assessment of left ventricular ejection fraction in critically ill patients: a bedside evaluation by novices and experts in echocardiography. Crit Care. 2022 Dec 14;26(1):386. doi: 10.1186/s13054-022-04269-6. PMID 36517906